CLINICAL TRIAL: NCT00300235
Title: The Epidemiology of Priapism (Sickle Cell Disease)
Brief Title: Priapism in Boys and Men With Sickle Cell Disease - Demographics, Characteristics and Prevalence
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Zora R. Rogers, Professor of Pediatrics, University of Texas Southwestern Medical Center
Other Study IDs: 1319; U54HL070587 (NIH)
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Priapism; Anemia, Sickle Cell
Keywords: Sickle Cell Anemia
MeSH Terms: conditions — Priapism; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- 1: 200 subjects ages 5 to 9.9 years with a diagnosis of HbSS/HbSβ0
- 2: 400 subjects ages 10 to 14.9 years with a diagnosis of HbSS/HbSβ0
- 3: 400 subjects ages 15 to 24.9 years with a diagnosis of HbSS/HbSβ0
- 4: 400 subjects over the age of 25 with a diagnosis of HbSS/HbSβ0
- 5: 250 subjects age 15 and older with a diagnosis of HbSC or HbSβ+

SUMMARY:
Priapism, a prolonged erection of the penis, is a medical issue that often affects men with sickle cell disease. The purpose of this study is to collect demographic and clinical information on priapism by interviewing men with sickle cell disease.

DETAILED DESCRIPTION:
Priapism is a prolonged, painful erection of the penis that lasts for more than four hours and occurs without sexual stimulation. It occurs when blood in the penis becomes trapped and is unable to drain properly. If it is not treated immediately, it can lead to scarring and permanent erectile dysfunction. Many cases of priapism are the result of sickle cell disease; approximately 42% of all adults with sickle cell disease will eventually develop priapism. Current treatments include medication, ice packs, or surgery. More research is needed to better understand the demographic and clinical characteristics of priapism. The purpose of this study is to collect information and further characterize priapism by conducting interviews with men with sickle cell disease. In turn, these findings may guide future priapism clinical trials.

This study will consist of two standardized questionnaires that will be administered to 1,650 men with sickle cell disease. Participants will complete an initial five-item questionnaire about priapism. If a participant indicates past experience with priapism on this initial questionnaire, he will be asked to complete a second questionnaire. This questionnaire will ask in-depth questions to further characterize the participant's episodes of priapism. If health issues such as drug use, harmful sexual behaviors, or impotence are identified upon reviewing the questionnaire, clinic staff will suggest care options and provide appropriate referrals to the participants. All participants will receive an educational brochure about priapism and compensation for completing the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell anemia or sickle beta zero thalassemia, if 5 years of age or over OR
* Diagnosis of sickle beta plus thalassemia or sickle hemoglobin C disease, if 15 years of age or over
* Participant and/or parent or guardian must be able to communicate adequately with the interviewer
* May participate if currently taking hydroxyurea, undergoing chronic transfusion, or participating in other research studies, including those involving treatments such as arginine, if all other inclusion criteria are met

Exclusion Criteria

Subjects who meet any of the following criteria are disqualified from enrollment in the study:

1. Patient or parent/guardian declines participation.
2. Female.
3. Subject or parent/guardian unable to communicate adequately with the interviewer.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males receiving care in any Comprehensive Sickle Cell Center.
Sampling Method: Non-Probability Sample
Enrollment: 1464 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Ballas, MD, Study Chair — Thomas Jefferson University; Lennette Benjamin, Study Chair — Montefiore Medical Center and Children's Hospital of Montefiore; J. Bessman, MD, Study Chair — University of Texas Southwestern at Galveston; Joan Cain, MD, Study Chair — UT Children's Hospital of Oklahoma; Lewis Hsu, MD, Study Chair — St. Christopher's Hospital; Laura DeCastro, MD, Study Chair — Duke University; Cage Johnson, MD, Study Chair — University of Southern California Los Angeles County & University of Southern California Medical Center; Karen Kalinyak, MD, Study Chair — Children's Hospital Medical Center, Cincinnati; Susan Lieff, PhD, Study Chair — Rho, Inc.; Lillian McMahon, MD, Study Chair — Boston Medical Center; William Mentzer, MD, Study Chair — University of California San Francisco Pediatric Hematology/Oncology; Ashok Raj, MD, Study Chair — Norton Healthcare; Rupa Redding-Lallinger, MD, Study Chair — University of North Carolina, Chapel Hill; Zora R. Rogers, MD, Study Chair — University of Texas Southwestern Medical Center at Dallas and Children's Medical Center; Cynthia Rutherford, MD, Study Chair — University of Texas, Southwestern Medical Center at Dallas; Kim Smith-Whitley, MD, Study Chair — Children's Hospital of Philadelphia; Elliott Vichinsky, MD, Study Chair — Children's Hospital and Research Center at Oakland & Summit Medical Center; Winfred Wang, MD, Study Chair — St. Jude Children's Research Hospital; Richard Snyder, MD, Study Chair — University of Cincinnati; Kathryn Hassell, MD, Study Chair — University of Colorado, Denver; Matthew Heeney, MD, Study Chair — Boston Children's Hospital; Eric Kraut, MD, Study Chair — Ohio State University; Stacy Month, MD, Study Chair — Kaiser Permanente - Oakland; Maureen Okam, MD, Study Chair — Dana-Farber Cancer Institute; Courtney Thornburg, MD, Study Chair — Duke University
Locations (27):
- United States (27):
  - University of South Alabama, Mobile, Alabama
  - University of California, Davis, Davis, California
  - Children's Hospital and Research Center at Oakland & Summit Medical Center, Oakland, California
  - Kaiser Permanente, Oakland, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Kosair Children's Hospital, Louisville, Kentucky
  - Brigham and Women's Hospital at Harvard Medical School, Boston, Massachusetts
  - Children's Hospital of Boston, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Children's Hospital Montefiore, The Bronx, New York
  - Montefiore Medical Center and Children's Hospital at Montefiore, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - St. Jude Children's Hospital, Memphis, Tennessee
  - University of Texas Parkland Health & Hospital System, Dallas, Texas
  - University of Texas Children's Medical Center of Dallas, Dallas, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Data still in analysis with NO FUNDING and all on paper from closure of contracted SDMC

RESULTS

PARTICIPANT FLOW:
Groups:
- Age 5-9.9 HbSS/HbSβ0: Subjects 5 to 9.9 yrs w/SCD diagnosis HbSS/HbSβ0
- Age 10-14.9 HbSS/HbSβ0: Subjects 10 to 14.9 ys w/SCD diagnosis HbSS/HbSβ0
- Age 15-24.9 HbSS/HbSβ0: Subjects 15 to 24.9 yrs w/SCD diagnosis HbSS/HbSβ0
- Age >25 HbSS/HbSβ0: Subjects > 25 yrs w/SCD diagnosis HbSS/HbSβ0
- Age >15 HbSC/HbSβ+: Subjects > 15 yrs w/SCD diagnosis HbSC/HbSβ+
Period: Overall Study
Arm/Group | Age 5-9.9 HbSS/HbSβ0 | Age 10-14.9 HbSS/HbSβ0 | Age 15-24.9 HbSS/HbSβ0 | Age >25 HbSS/HbSβ0 | Age >15 HbSC/HbSβ+
Started | 208 | 240 | 398 | 362 | 251
Completed | 208 | 240 | 398 | 362 | 251
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 5-9.9 HbSS/HbSβ0 | Age 10-14.9 HbSS/HbSβ0 | Age 15-24.9 HbSS/HbSβ0 | Age >25 HbSS/HbSβ0 | Age >15 HbSC/HbSβ+ | Total
Number analyzed (Participants) | 208 | 240 | 398 | 362 | 251 | 1459
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 208 | 240 | 203 | 0 | 84 | 735
  Between 18 and 65 years | 0 | 0 | 195 | 361 | 165 | 721
  >=65 years | 0 | 0 | 0 | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.4 (1.44) | 12.6 (1.46) | 19.3 (2.72) | 36.0 (8.93) | 29.8 (13.69) | 22.5 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 208 | 240 | 398 | 362 | 251 | 1459
Region of Enrollment [Number; unit: participants]
  United States | 208 | 240 | 398 | 362 | 251 | 1459.0

OUTCOME MEASURES:

1. Primary Outcome: Enumeration of the Prevalence of Priapism in Males With Sickle Cell Anemia and Sickle Beta Zero Thalassemia.
Description: Subject responded YES to survey Question "Have you ever had priapism?". By diagnosis and age group. Enumeration of the prevalence of priapism in males with sickle cell anemia and sickle beta zero thalassemia.
Time Frame: At time of interview
Population: All particpants who completed survey were analyzed.
Measure: Number; unit: participants
Arm/Group | Age 5-9.9 HbSS/HbSβ0 | Age 10-14.9 HbSS/HbSβ0 | Age 15-24.9 HbSS/HbSβ0 | Age >25 HbSS/HbSβ0 | Age >15 HbSC/HbSβ+
Number analyzed (Participants) | 208 | 240 | 398 | 362 | 251
participants | 18 | 58 | 160 | 189 | 60
Statistical Analysis 1: Comparison: Age 5-9.9 HbSS/HbSβ0; This was a survey designed to estimate prevalence, no formal comparisons between age or genotype groups were performed; Test type: Superiority or Other; proportion of subjects = 35.2, 95% CI [32.5 to 37.9]

2. Secondary Outcome: Characterization of Priapism in Males With Sickle Cell Anemia With Reference to Time of Onset, Duration of Events, Frequency of Episodes, Precipitating or Associated Activities, Treatment Modalities Used, and Outcome of Treatments
Description: Characterization of priapism in males with sickle cell anemia with reference to time of onset, duration of events, frequency of episodes, precipitating or associated activities, treatment modalities used, and outcome of treatments.
Time Frame: Cross-sectional single survey visit
Reporting Status: Not Posted

3. Secondary Outcome: Descriptive Comparison of the Prevalence of Priapism in Males With Sickle Cell Anemia to That Described in Older Patients With Other Sickle Hemoglobinopathies
Description: Descriptive comparison of the prevalence of priapism in males with sickle cell anemia to that described in older patients with other sickle hemoglobinopathies.
Time Frame: Cross-sectional single survey visit
Reporting Status: Not Posted

4. Secondary Outcome: Assessment of General Patient and Parent Understanding of Priapism as a Complication of Sickle Cell Disease Gained From Completion of Protocol
Description: Assessment of general patient and parent understanding of priapism as a complication of sickle cell disease gained from completion of protocol.
Time Frame: Cross-sectional single survey visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Age 5-9.9 HbSS/HbSβ0 | Age 10-14.9 HbSS/HbSβ0 | Age 15-24.9 HbSS/HbSβ0 | Age >25 HbSS/HbSβ0 | Age >15 HbSC/HbSβ+
Serious Adverse Events (participants affected / at risk) | 0/208 | 0/240 | 0/398 | 0/362 | 0/251
Other Adverse Events (participants affected / at risk) | 0/208 | 0/240 | 0/398 | 0/362 | 0/251

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No